CLINICAL TRIAL: NCT05398965
Title: Eucalyptus Oil as Adjuvant Therapy for Coronavirus Disease 19 (COVID-19), a Randomized Open-label Clinical Trial
Brief Title: Eucalyptus Oil as Adjuvant Therapy for Coronavirus Disease 19 (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hasanuddin University (Other)
Collaborators: Ministry of Agriculture, Republic of Indonesia (Unknown)
Responsible Party: Principal Investigator, Bumi Herman, Assistant Lecturer, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3105221321
Record Dates: First submitted 2022-05-31; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: COVID-19; Eucalyptus; Viral Clearance; Cytokine Level; Clinical Improvement
MeSH Terms: conditions — COVID-19 | interventions — Eucalyptus Oil

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into 2 study groups before starting their medication. The first group was only given standard COVID-19 therapy. While the treated group will be given standard COVID-19 along with adjuvant therapy (Eucalyptus oil on external use)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The group will receive standard COVID medication + Eucalyptus oil on external use for 14 days
  Interventions: Drug: Eucalyptus Oil; Drug: Standard COVID medication
- Comparator Group (Active Comparator): The group will receive standard COVID medication only
  Interventions: Drug: Standard COVID medication

INTERVENTIONS:
Drug: Eucalyptus Oil — The Eucalyptus Oil pack contains Oleum Eucalyptus citriodora, Oleum Eucalyptus globulus, and Peppermint oil, given 4 times daily for 45 minutes each frequency, applied to the mask.
  Other Names: Herbal Roll On
  Arms: Intervention Group
Drug: Standard COVID medication — This standard treatment is personalized according to the severity but is not limited to standard antiviral therapy, azithromycin 500 mg a day, vitamin C 500 mg 8 hourly a day, zinc 20 mg a day, tablet of complex vitamin B, and other symptomatic treatments.
  Other Names: COVID Medication

SUMMARY:
Background :

Based on several clinical trials, eucalyptus oil can suppress edema formation and reduce inflammation, where the effect of 1,8-cineole is due to the inhibition of cytokine secretion by T lymphocytes. This but not limited to the reduction of interleukin (IL) of IL-4, IL-5, and IL-10 in nasal lavage fluids and levels of IL- 1β, IL-6, Tumor Necrosis Factor-α (TNF-α), and Interferon-γ (IFN-γ) in lung tissue of mice infected with influenza virus. Hence the researchers assume that Eucalyptus may possess benefits in COVID-19 as adjuvant therapy.

Objectives :

The primary objective of this study is to evaluate the efficacy of Eucalyptus oil as adjuvant therapy in mild-moderate COVID-19 patients.

Hypothesis :

Eucalyptus oil may reduce the inflammatory cytokines which eventually improves clinical symptoms

DETAILED DESCRIPTION:
Detailed Objectives :

1. To assess the safety of Eucalyptus oil as an adjuvant to the standard of care in treating patients with mild to moderate COVID-19 symptoms.
2. To document the effect of Eucalyptus oil on clinical symptoms improvement, including cough, anosmia, and sore throat.
3. To assess the effect of Eucalyptus oil on viral load indirectly reflected by the Real Time-Polymerase Chain Reaction/RT-PCR cycle threshold (CT)
4. To assess the effect of Eucalyptus oil on NLR, Interleukin-6, Interleukin-10, and Tumor Growth Factor-β (TGF-β) as inflammatory marker
5. To assess the effect of Eucalyptus oil on immunoglobulin (Ig) M and G in patient's serum

Target population:

Patients with mild-moderate COVID-19

Setting:

Hospital and outpatient care

Intervention:

External use of Eucalyptus oil

Subject Recruitment and Screening :

1. A written, signed, and dated (ICF) consent form will be obtained from the patient before the study's inclusion. Assessment and records of patient's clinical report forms including demographic data, comorbidities and concurrent medications, symptoms experienced by the patient, body weight, height of the body, body mass index, vital signs, and fingertip oxygen saturation.
2. Baseline laboratory tests including complete blood count (CBC), neutrophil-lymphocyte ratio (NLR), liver (alanine aminotransferase (ALT), aspartate aminotransferase (AST), kidney function tests (serum creatinine), serum ferritin, blood glucose, coagulation test (prothrombin time and activated partial thromboplastin time), cytokine level (IL-6, IL-10, and TGF-β) will be assessed. On admission, computed tomography (CT) scan of the chest will also be performed.

Detailed procedures :

Eucalyptus oil will be applied to the surgery mask, 4 times a day, which is 45 minutes duration in each session for 14 days. Clinical assessment and vital signs, and follow-up RT-PCR tests by nasopharyngeal swab will be documented on days 5, 10, and 15. Follow-up laboratory results for blood, liver function, kidney function, blood glucose, cytokine level, and CT scan will be performed on Day 15. If moderate COVID-19 patients confirmed negative RT-PCR test results in 2 consecutive tests, the patient is allowed to be discharged and continue their adjuvant treatment at home (in the intervention group).

Sample size estimation :

following the sample size estimation of two different means

1. Type 1 error 5%
2. Power of study 80%
3. superiority trial hypothesis
4. equal allocation for two arms

f. effect size is estimated at 0.7 total sample required : 52

Statistical Analysis

1. Intention to treat
2. Descriptive statistic
3. Repeated measurement analysis using mixed model analysis.

ELIGIBILITY:
Inclusion Criteria:

1. SARS-COV-2 infections were confirmed by real-time reverse transcription-polymerase chain reaction (RT-PCR) from the nasopharyngeal swab.
2. Mild to moderate clinical symptoms or with nasal cannula oxygen modality maximal oxygen 4 liters/minute (Moderate COVID-19 patients mean patients with clinical signs of pneumonia (fever, cough, shortness of breath, rapid breathing) but no signs of severe pneumonia including Oxygen Saturation ≥ 95%)
3. Sign the informed consent
4. Have not received the COVID-19 medicine yet

Exclusion Criteria:

1. They have or develop severe COVID-19 symptoms according to the COVID-19 diagnosis and treatment guidelines of Indonesian society of respiratory; respiratory distress (RR ≥30 breaths/min, oxygen saturation <95% at a rest state)
2. History of hepatitis or impaired liver function
3. Patients with or had a history of comorbid such as coronary heart disease, congestive heart disease, renal insufficiency, chronic liver disease, diabetes mellitus, uncontrolled hypertension or grade II hypertension or hypertensive crisis, immunocompromised, Central Nervous System disorders (such as stroke, epilepsy, Alzheimer's, and meningitis)
4. Pregnant or lactating women
5. Allergy to any of the components of the test product
6. Participated in other clinical studies

Withdraw from the study:

The protocol treatment will be discontinued if the patient

1. Withdraw their consent based on the patient's demand
2. Patient's compliance of the use of test product <90% or >5 times not using the product according to the predetermined schedule
3. Severe adverse events occurred
4. After undergoing clinical trials, the patient experienced things that caused him/her to no longer meet the criteria set out in this protocol.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Clinical Symptoms | change of score for each symptoms from baseline to day 15
  The patient will be asked for clinical improvement (three symptoms, sore throat, anosmia and cough) with a 6-likert scale question for each symptoms. Higher number (5) indicates very severe symptoms whereas 0 indicates no symptoms.
Viral clearance | change of CT Value from baseline to day 15
  level of Severe Acute Respiratory Corona Virus 2 (SARS-COV2) on nasopharyngeal sample measured by RT-PCR in Cycle Threshold Unit (CT)
Neutrophil-Lymphocyte Ratio (NLR) | change of NLR from baseline to day 15
  This ratio is used as a marker of subclinical inflammation. It is calculated by dividing the number of neutrophils by number of lymphocytes from the blood sample

SECONDARY OUTCOMES:
Radiology improvement | change of radiology feature from baseline to day 15
  the Radiology improvement of lung Computed Tomography (CT-Scan) on day 15 indicates by resolution or absence of inflammatory sign or abnormal findings (binary response)
Cytokine level | change of cytokine level from baseline to day 15
  reduction of pro-inflammatory cytokine level in blood samples (Interleukin-6, Interleukin-10, Tumor Growth Factor/TGF-β)

CONTACTS AND LOCATIONS:
Overall Officials: Arif Santoso, MD, Ph.D, Principal Investigator — Hasanuddin University; Idrus Paturusi, Prof., Principal Investigator — Hasanuddin University; Nasrum Massi, Prof., Principal Investigator — Hasanuddin University; Idrianti Idrus, MD, Principal Investigator — Hasanuddin University; Firdaus Hamid, MD. PhD, Principal Investigator — Hasanuddin University; Andi Rofian Sultan, MD. Ph.D, Principal Investigator — Hasanuddin University; Munawir Munawir, MD, Principal Investigator — Hasanuddin University; Rasiha Rasiha, Principal Investigator — Hasanuddin University
Locations (1):
- Hasanuddin University Hospital, Makassar, South Sulawesi, Indonesia